CLINICAL TRIAL: NCT05288816
Title: A Phase 1, Open-Label, Single Ascending and Multiple Set Dose Study to Evaluate the Safety, Tolerability, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of ALXN1210 Administered Intravenously to Healthy Japanese Subjects
Brief Title: A Study of Single and Multiple Doses of ALXN1210 in Healthy, Adult Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ALXN1210-HV-104; 2015-005468-40 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: ALXN1210; Pharmacokinetics; Pharmacodynamics; Safety; Immunogenicity
MeSH Terms: interventions — ravulizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: ALXN1210 400 mg (Single) (Experimental): A single dose of ALXN1210 was administered intravenously.
  Interventions: Drug: ALXN1210
- Cohort 2: ALXN1210 800 mg (Single) (Experimental): A single dose of ALXN1210 was administered intravenously.
  Interventions: Drug: ALXN1210
- Cohort 3: ALXN1210 800 mg (Multiple) (Experimental): ALXN1210 (800 mg) was administered intravenously every 4 weeks for a total of 5 doses.
  Interventions: Drug: ALXN1210

INTERVENTIONS:
Drug: ALXN1210 — Participants received a single dose (400 mg or 800 mg) and multiple doses (800 mg) of ALXN1210.
  Other Names: Ultomiris; Ravulizumab

SUMMARY:
This study evaluated the safety and tolerability of single and multiple doses (400 and 800 milligrams [mg]) of ALXN1210 following intravenous administration to healthy Japanese participants.

DETAILED DESCRIPTION:
A total of 3 cohorts were enrolled sequentially. Participants received different doses per Cohorts: Cohort 1, 400 mg single dose; Cohort 2, 800 mg single dose; and Cohort 3, 800 mg every 4 weeks for a total of 5 doses. The Safety Review Committee (SRC) conducted a review of the available clinical and safety data after the last participants in the 400 mg cohort (Cohort 1) completed Day 15 to determine if dose escalation to the single dose 800 mg (Cohort 2) could proceed. The SRC then conducted a review of all available clinical and safety data after the last participants in Cohort 2 completed Day 15 to determine if dosing of Cohort 3 could begin. A 120-day (Cohort 1) or 140-day (Cohort 2) Follow-up Period was performed for safety, pharmacokinetic (PK), pharmacodynamic (PD), and immunogenicity assessments. Participants in Cohort 3, however, had a 185-day Follow-up Period for safety, PK, PD, and immunogenicity assessments after the fifth dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese males or females aged 25 through 55 years, inclusive (participants who lived outside of Japan for ≤ 10 years and were first-generation Japanese, defined as born in Japan and having 4 biological grandparents who were ethnic Japanese).
* Body mass index from 18 through 29.9 kilogram/square meter (kg/m^2), inclusive, with weight between 50 and 100 kg, inclusive.
* QT interval (corrected using the Fridericia's formula) ≤ 450 milliseconds (msec) for males and ≤ 470 msec for females at Screening and prior to dosing on Day 1.
* Willing and able to give written informed consent and comply with the study visit schedule
* Documented vaccination with tetravalent meningococcal conjugate vaccine (MCV4) at least 56 days and not more than 3 years prior to dosing. Documentation included a positive serum bactericidal assay to confirm an immune response before study drug administration.
* Vaccination with serogroup B meningococcal vaccine at least 56 days prior to dosing on Day 1, with a booster administered at least 28 days prior to dosing on Day 1, with at least 28 days between the first and second injections.
* Female participants of childbearing potential were required to use highly effective contraception, starting at Screening and continuing until at least 6 months (Cohort 1) or 8 months (Cohorts 2 and 3) after the last dose of ALXN1210.
* Male participants with a female spouse/partner of childbearing potential or a pregnant or breastfeeding spouse or partner had to agree to use barrier contraception during the treatment period and for at least 6 months (Cohort 1) or 8 months (Cohorts 2 and 3) after the last dose of ALXN1210.

Exclusion Criteria:

* Participants who were in intimate and prolonged contact with (defined as living under the same roof or providing personal care) people younger than 2 years of age or older than 65 years of age, or who were either immunocompromised or had one of the following underlying medical conditions: anatomic or functional asplenia (including sickle cell disease); congenital complement, properdin, factor D, or primary antibody deficiencies; acquired complement deficiencies (for example, those receiving eculizumab); or human immunodeficiency virus (HIV).
* Participants who were professionals exposed to environments of greater risk for meningococcal disease; research, industrial, and clinical laboratory personnel routinely exposed to Neisseria meningitidis; military personnel during recruit training (military personnel may be at increased risk of meningococcal infection when accommodated in close quarters); daycare center workers; those who lived on a college or university campus; and those who planned to travel during the course of the study or have travelled to endemic areas for meningococcal meningitis (for example, India, Sub-Saharan Africa, pilgrimage to Saudi Arabia for Hajj) 6 months prior to dosing.
* History of any Neisseria infection
* History of unexplained, recurrent infection; or infection requiring treatment with systemic antibiotics within the 90 days prior to dosing.
* HIV infection (evidenced by HIV-1 or HIV-2 antibody titer)
* Acute or chronic hepatitis B virus infection. Hepatitis B surface antigen (HBsAg) testing was required for all participants prior to enrollment. Participants with positive HBsAg were not enrolled. For participants with negative HBsAg, the following testing algorithms were required: If hepatitis B core antibody (HBcAb) was negative, the participants was eligible to enroll and If HBcAb was positive, the hepatitis B surface antibody (HBsAb) was tested. (If both HBcAb and HBsAb were positive, the participants was eligible to enroll and If HBcAb was positive and HBsAb was negative, the participants was not enrolled.)
* Acute or chronic hepatitis C virus infection (evidenced by antibody titer)
* Active systemic viral or fungal infection 14 days prior to dosing.
* Positive or indeterminate QuantiFERON-TB test indicating possible tuberculosis infection.
* History of latent or active tuberculosis or exposure to endemic areas within 8 weeks prior to the Screening Visit.
* Female participants who were breastfeeding or were unwilling to practice contraception and were not postmenopausal.
* Positive serum pregnancy test at Screening or Day -1.
* Serum creatinine greater than the upper limit of normal (ULN) of the reference range of the testing laboratory at Screening or Day -1.
* Alanine aminotransferase or aspartate aminotransferase > ULN of the reference range of the testing laboratory at Screening or > 1.5*ULN of the reference range of the testing laboratory at Day -1.
* Any of the following hematology results: hemoglobin < 130 grams (g)/L for males and < 115 g/L for females; hematocrit < 0.37 L/L for males and < 0.33 L/L for females; white blood cells < 3.0*10^3/microliter (μL); absolute neutrophils < 2.0*10^3/μL; and platelets < 150 or > 400*10^3/μL at Screening or Day -1; or complete blood count clinical laboratory results that were considered clinically relevant and unacceptable by the investigator at Day -1.
* History of complement deficiency or complement activity below normal reference range as evaluated by complement alternative pathway enzyme-linked immunosorbent assay at Screening.
* History of malignancy with the exception of a nonmelanoma skin cancer or carcinoma in situ of the cervix that had been treated with no evidence of recurrence.
* Participated in a clinical study within 30 days before initiation of dosing on Day 1 or use of any experimental small-molecule therapy within 30 days prior to dosing on Day 1.
* Participated in more than 1 clinical study of a monoclonal antibody (mAb), or participation in a clinical study of an mAb within the 12 months prior to Screening, during which the participants was exposed to the active study drug. Participants who participated in only 1 study of an mAb could have been considered for enrollment if they completed that study more than 12 months prior to Screening.
* Major surgery or hospitalization within 90 days prior to dosing.
* Contraindication to receiving MCV4 and/or serogroup B vaccine, including severe allergic reaction to a previous dose of MCV4 and/or serogroup B vaccine; severe allergy to any vaccine component; or previous diagnosis of Guillain-Barré syndrome.
* History of allergy to excipients of ALXN1210 (for example, polysorbate 80)
* Documented history of penicillin or cephalosporin
* History of significant allergic reaction (anaphylaxis, or angioedema) to any product (for example, food and pharmaceutical).
* Smoked > 10 cigarettes daily (former smokers may have been permitted to enroll at the Investigator's discretion)
* Positive urine drug toxicology screen at Screening or Day -1.
* Donated plasma within 7 days prior to dosing. Donated or lost more than 50 mL of blood within 30 days of dosing or lost more than 499 mL of blood within 56 days of dosing
* Used prescription medications within 14 days prior to study drug administration.
* Clinical diagnosis of any autoimmune or rheumatologic disease.
* Immunized with a live-attenuated vaccine 1 month prior to dosing or planned vaccination during the course of the study (except for the vaccination planned by the study protocol). Immunization with inactivated or recombinant influenza vaccine was permitted.
* Had fever (confirmed body temperature > 37.6°C) (for example, a fever associated with a symptomatic viral or bacterial infection) within 14 days prior to the first dosing.
* Participants with any medical history, conditions or risks which, in the opinion of the Investigator, may have interfered with the participant's full participation in the study, or compliance with the protocol, or posed any additional risk for the participant, or confounded the assessment of the participant or outcome of the study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-18 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: ALXN1210 400 mg Single Dose: Participants received a single dose of ALXN1210 400 milligrams (mg), via intravenous (IV) infusion on Day 1. Participants were followed for 120 days.
- Cohort 2: ALXN1210 800 mg Single Dose: Participants received a single dose of ALXN1210 800 mg, via IV infusion on Day 1. Participants were followed for 140 days.
- Cohort 3: ALXN1210 800 mg Multiple Dose: Participants received multiple doses of ALXN1210 800 mg, via IV infusion every 4 weeks (on Days 1, 29, 57, 85, and 113) for a total of 5 doses. Participants were followed for 185 days.
Period: Overall Study
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose | Cohort 3: ALXN1210 800 mg Multiple Dose
Started | 4 | 4 | 8
Received at Least 1 Dose of Study Drug | 4 | 4 | 8
Completed | 4 | 4 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Groups:
- Cohort 1: ALXN1210 400 mg Single Dose: Participants received a single dose of ALXN1210 400 mg, via IV infusion on Day 1. Participants were followed for 120 days.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose | Cohort 3: ALXN1210 800 mg Multiple Dose | Total
Number analyzed (Participants) | 4 | 4 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (7.32) | 35.0 (8.72) | 30.9 (4.32) | 32.4 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 2 | 0 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 4 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign (for example, including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product or procedure, whether or not considered related to the medicinal product or procedure, which occurred during the course of the clinical study. TEAEs were defined as AEs that occurred on or after the date and time of study drug administration, or those that first occurred before dosing but worsened in frequency or severity after study drug administration. A summary of all Serious Adverse Events and Other Adverse Events (nonserious) regardless of causality is located in the 'Reported Adverse Events' Section.
Time Frame: Cohort 1: Baseline up to Day 120; Cohort 2: Baseline up to Day 140; Cohort 3: Baseline up to Day 298
Population: The safety population consisted of all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 4 | 4 | 8
Participants | 2 | 3 | 8

2. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) To ALXN1210
Description: Blood samples were collected to evaluate antibody response through development of ADAs.
Time Frame: Cohort 1: Baseline up to Day 120; Cohort 2: Baseline up to Day 140; Cohort 3: Baseline up to Day 298
Population: The immunogenicity analysis population consisted of all participants who had a pre-dose and post-dose ADA samples collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 4 | 4 | 8
Participants | 0 | 0 | 0

3. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero To Infinity (AUCinf) For Single Dose of ALXN1210
Description: Blood samples were collected for estimation of AUCinf using Phoenix WinNonlin software version 7.0.
Time Frame: Cohort 1: Baseline (pre-dose) up to Day 120; Cohort 2: Baseline (pre-dose) up to Day 140
Population: The pharmacokinetic (PK) population consisted of all participants who had sufficient serum concentration data to enable the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: hour*microgram/milliliter (hr*mcg/mL)
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose
Number analyzed (Participants) | 4 | 4
hour*microgram/milliliter (hr*mcg/mL) | 102361.591 (22918.174) | 261313.227 (16016.673)

4. Secondary Outcome: Area Under The Serum Concentration Versus Time Curve From Time Zero To Infinity (AUCinf) For Multiple Dose of ALXN1210
Description: Blood samples were collected for estimation of AUCinf using Phoenix WinNonlin software version 7.0.
Time Frame: Day 113 (pre-dose) up to Day 298
Population: The PK population consisted of all participants who had sufficient serum concentration data to enable the calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: hr*mcg/mL
Arm/Group | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 8
hr*mcg/mL | 499626.032 (116203.665)

5. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) For Single Dose of ALXN1210
Description: Blood samples were collected for estimation of Cmax using Phoenix WinNonlin software version 7.0.
Time Frame: Cohort 1: Baseline (pre-dose) up to Day 120; Cohort 2: Baseline (pre-dose) up to Day 140
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose
Number analyzed (Participants) | 4 | 4
micrograms/milliliter | 174.750 (25.316) | 397.750 (25.526)

6. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) For Multiple Dose of ALXN1210
Description: Blood samples were collected for estimation of Cmax using Phoenix WinNonlin software version 7.0.
Time Frame: Day 113 (pre-dose) up to Day 298
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 8
mcg/mL | 565.625 (76.651)

7. Secondary Outcome: Percent Change From Baseline in Free Complement Protein C5 Concentration at Day 1
Time Frame: Baseline, Day 1 (end of infusion)
Population: The pharmacodynamic (PD) population consisted of all participants who had sufficient total and free C5 concentration data and chicken red blood cells (cRBC) hemolysis data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose
Number analyzed (Participants) | 4 | 4
percent change | -99.7762 (0.0617) | -99.8920 (0.0333)

8. Secondary Outcome: Percent Change From Baseline in Free Complement Protein C5 Concentration at Day 113
Time Frame: Baseline, Day 113 (end of infusion)
Population: The PD population consisted of all participants who had sufficient total and free C5 concentration data and cRBC hemolysis data.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 8
percent change | -99.5724 (0.0492)

9. Secondary Outcome: Percent Change From Baseline in Total C5 Concentration at Day 1
Time Frame: Baseline, Day 1 (end of infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose
Number analyzed (Participants) | 4 | 4
percent change | -5.0810 (4.7737) | -5.5713 (2.6475)

10. Secondary Outcome: Percent Change From Baseline in Total C5 Concentration at Day 113
Time Frame: Baseline, Day 113 (end of infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 8
percent change | -8.3487 (3.5507)

11. Secondary Outcome: Percent Change From Baseline in Chicken Red Blood Cell Hemolysis at Day 1
Time Frame: Baseline, Day 1 (end of infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose
Number analyzed (Participants) | 4 | 4
percent change | -98.9905 (1.8232) | -98.5454 (2.2934)

12. Secondary Outcome: Percent Change From Baseline in Chicken Red Blood Cell Hemolysis at Day 113
Time Frame: Baseline, Day 113 (end of infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Cohort 3: ALXN1210 800 mg Multiple Dose
Number analyzed (Participants) | 8
percent change | -97.8156 (2.9408)

ADVERSE EVENTS:
Time Frame: Cohort 1: Baseline up to Day 120; Cohort 2: Baseline up to Day 140; Cohort 3: Baseline up to Day 298
Description: The safety population consisted of all participants who received at least 1 dose of study drug.
Arm/Group | Cohort 1: ALXN1210 400 mg Single Dose | Cohort 2: ALXN1210 800 mg Single Dose | Cohort 3: ALXN1210 800 mg Multiple Dose
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 2/4 | 3/4 | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: ALXN1210 400 mg Single Dose (N=4) | Cohort 2: ALXN1210 800 mg Single Dose (N=4) | Cohort 3: ALXN1210 800 mg Multiple Dose (N=8)
Eyelids pruritus (Eye disorders) | 0 | 1 | 0
Photopsia (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1
Libido decreased (Psychiatric disorders) | 0 | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT05288816/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT05288816/SAP_001.pdf